CLINICAL TRIAL: NCT04622982
Title: Efficacy and Safety of a Long-term Multidisciplinary Weight Loss Intervention in Patients With Obesity: an Open Label Study
Brief Title: A Multidisciplinary Intervention for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206/151217
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Vitamin D; Exercise; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Open Label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Obese subjects with BMI >= 30 and with one or more of metabolic comorbidities (type 2 diabetes mellitus, dyslipidemia, high blood pressure, hyperuricemia, and others).
  Interventions: Other: Multidisciplinary treatment of obesity (diet + vitamin D + exercise + psychotherapy)

INTERVENTIONS:
Other: Multidisciplinary treatment of obesity (diet + vitamin D + exercise + psychotherapy) — Body weight reduction was induced by a low-energy mixed diet (55 % carbohydrates, 30 % lipids and 15 % proteins) providing 600 kcal less than individually estimated energy requirements based on the measured REE. The energy content and macronutrient composition of the diets adhered to the nutritional recommendations of the American Diabetes Association.
  Patients were administered vitamin D supplement only if they presented a value of 25-hydroxyvitamin D (25OHD) <30 ng/ml in blood tests at the beginning.
  Patients were following an individualized physical activity plan within the hospital and were aided by a psychodynamic approach therapist.

SUMMARY:
This is an open label study in which obese participants were treated with a restrictive hypo-caloric diet under hospitalization for a maximum period of 3 months in a metabolic rehabilitation unit. A multidisciplinary approach was used (combination of diet, physical exercise and psychotherapy)

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* BMI >= 30
* one or more comorbidities (type 2 diabetes mellitus, dyslipidemia, high blood pressure, hyperuricemia, and others)

Exclusion Criteria:

* active cancer
* severe cognitive or functional impairments
* severe behavioral disorders
* known kidney failure (previous glomerular filtration rate <30 ml/min)
* known liver failure (Child B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
  Change in body Weight

SECONDARY OUTCOMES:
GlycaemIa | 12 weeks
  Change in glycaemia
Insulin | 12 weeks
  Change in insulin blood levels
Homa IR | 12 weeks
  Change in HOMA-IR
Total cholesterol | 12 weeks
  Change in blood total cholesterol
LDL cholesterol | 12 weeks
  Change in LDL cholesterol
HDL cholesterol | 12 weeks
  Change in HDL cholesterol
Triglycerides | 12 weeks
  Change in triglycerides
AST (Aspartate Aminotransferase) | 12 weeks
  Change in blood of Aspartate Aminotransferase (AST)
ALT (alanine aminotransferase) | 12 weeks
  Change in blood of alanine aminotransferase (ALT)
GGT (gamma-glutamyl transpeptidase) | 12 weeks
  Change in blood of gamma-glutamyl transpeptidase (GGT)
Total bilirubin | 12 weeks
  Change in blood total bilirubin
Basal metabolic rate | 12 weeks
  Change in basal metabolic rate

OTHER OUTCOMES:
Body composition - Body Fat Mass | 12 weeks
  Change in Body Fat
Body composition - Body Fat free mass | 12 weeks
  change in Body Fat free mass
Body composition - Visceral Fat mass | 12 weeks
  change in Visceral Fat mass
Body Circumferences - arm | 12 weeks
  change in circumferences (arm)
Body Circumferences - calf | 12 weeks
  change in circumferences (calf)
Body Circumferences - waist | 12 weeks
  change in circumferences ( waist)
Body Circumferences - hips | 12 weeks
  change in circumferences (hips)
Iron | 12 weeks
  Change in blood Iron concentration
Other biochemical parameters - vit D | 12 weeks
  Change in blood vitamin D
Other biochemical parameters - vit B12 | 12 weeks
  Change in blood vitamin B12
Other biochemical parameters - Folates | 12 weeks
  Change in blood Folates
Other biochemical parameters - transferrin | 12 weeks
  Change in transferrin
Other biochemical parameters - Homocystein | 12 weeks
  Change in Homocystein
Other biochemical parameters - albumin | 12 weeks
  Change in blood proteins (albumin)
Other biochemical parameters - prealbumin | 12 weeks
  Change in blood proteins (prealbumin)
Other biochemical parameters - enzymes - lipase | 12 weeks
  Change in blood enzymes (lipase)
Other biochemical parameters - enzymes - amylase | 12 weeks
  Change in blood enzymes (amylase)
Other biochemical parameters - thyroid hormones - FT3 | 12 weeks
  Change in FT3
Other biochemical parameters - thyroid hormones - FT4 | 12 weeks
  Change in FT4
Other biochemical parameters - thyroid hormones - TSH | 12 weeks
  Change in TSH
Other biochemical parameters - inflammatory markers - CRP | 12 weeks
  Change in C-reactive protein
Other biochemical parameters - inflammatory markers - ESR | 12 weeks
  Change in Erythrocyte Sedimentation Rate
Other biochemical parameters - creatinin | 12 weeks
  Change in blood creatinin
Uric acid | 12 weeks
  Change in uric acid blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, MD, PhD, Study Director — Azienda di Servizi alla Persona di Pavia

IPD SHARING:
Plan to Share IPD: No
IPD are not shared. Published article will display mean baseline values and mean differences from baseline.